CLINICAL TRIAL: NCT05819307
Title: Structural Imaging Assisted Retinal Fluorescence Lifetime Imager (STARFLI) Using a High-speed Fluorescence Lifetime Measurement Scheme
Brief Title: Structural Imaging Assisted Retinal Fluorescence Lifetime Imager (STARFLI)
Acronym: STARFLI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Haag-Streit AG (Industry); University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: STARFLI
Record Dates: First submitted 2023-03-01; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-03

CONDITIONS: Retinal Disease
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: OCT/FLIM — OCT/FLIM imaging of the retina

SUMMARY:
To investigate the feasibility of a combined OCT/FLIM device

DETAILED DESCRIPTION:
To investigate the feasibility of a combined Optical coherence tomography/ Fluorescence Lifetime Measurement (OCT/FLIM) device.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be willing to give written informed consent
* Age: Patients and Probands 18 years or greater
* Both eyes will be assessed in the study

Exclusion Criteria:

* Patients not willing or able to sign informed consent
* Patients younger than 18 years
* Patients with epilepsy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Retina healthy subjects
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of device | 1 year
  We will organize and perform an observational study with the prototype OCT+FLIM device and contribute the acquired OCT/FLIM datasets from eyes of different age and status of the crystalline lens.

SECONDARY OUTCOMES:
To provide two key technology aspects of the project: | 1 year
  A. The first will be to bring forward a novel registration strategy for calibrated OCT and FLIM modalities, so that these can be used in conjunction.
  B. The second will be to develop an image calibration and normalization method using the measured lens fluorescence lifetime and possibly also structural (OCT) information on lens and retina, so that data acquired by the device can be used across different patients in a consistent way.

CONTACTS AND LOCATIONS:
Overall Officials: Martin S. Zinkenagel, Prof.Dr.Dr., Study Chair — Clinic director
Locations (1):
- Department of Ophthalmology, Bern University Hospital, Bern, 3010 Bern, Switzerland, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No